CLINICAL TRIAL: NCT01820780
Title: Usefulness of a Short-time But Very Early Specialized Follow-up After Hospitalization for Acute Heart Failure: a Randomized Controlled Trial.
Brief Title: Early Care After Discharge of HF Patients
Acronym: ECAD-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110128
Record Dates: First submitted 2013-01-25; First posted 2013-03-29 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Disease management program
MeSH Terms: conditions — Heart Failure | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive disease management (Experimental): Planned consultations with HF specialist including biological test at weeks 1, 2 and 4; in addition to usual care.
  Interventions: Other: Natriuretic peptides levels to J7 and J14; Other: Consultations specialized to J7 and J14; Other: Phone calls in 6 months and 12 months; Other: Natriuretic peptides levels at 6 months; Other: Consultation with the general doctor or the cardiologist to J30 with blood results
- usual disease management (Active Comparator): usual care according to guidelines; including first medical consultation and biological test within the 4-week time following discharge.
  Interventions: Other: Phone calls in 6 months and 12 months; Other: Natriuretic peptides levels at 6 months; Other: Consultation with the general doctor or the cardiologist to J30 with blood results

INTERVENTIONS:
Other: Natriuretic peptides levels to J7 and J14
  Arms: intensive disease management
Other: Consultations specialized to J7 and J14 — Optimization of treatments Education on the signs of alert of the disease and on the medicines Reduction of the rate of BNP or NTproBNP = 30 % between the exit of the hospitalization and the second consultation Planning of an adapted coverage
  Arms: intensive disease management
Other: Phone calls in 6 months and 12 months
Other: Natriuretic peptides levels at 6 months
Other: Consultation with the general doctor or the cardiologist to J30 with blood results

SUMMARY:
After decompensated heart failure, a number of patients have high risk of early rehospitalization as well as death. Specialized medical management for a short period but very early after discharge could be critical for optimizing care and improving early outcome.

This study aims to compare such early intensive medical management with usual care in high-risk patients after discharge.

DETAILED DESCRIPTION:
At discharge, high-risk HF patients are selected and randomized in two groups:

* Control group: usual disease management according to guidelines and including first medical consultation and biological test within the 4-week time following discharge.
* Active group: consultations with HF specialist including biological test at weeks 1, 2 and 4 are planned in addition to usual management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* consent signed
* Acute or decompensated heart failure with one or more of following criteria::

  * Discharge BNP > 350 pg/ml or NTproBNP > 2200 pg/ml
  * Discharge serum creatinine ≥ 180µM
  * Discharge systolic blood pressure ≤ 110mmHg
  * Previous hospitalisation for acute heart failure < 6 months

Exclusion Criteria:

* acute coronary syndrome,
* acute myocarditis,
* isolated right HF,
* transient HF,
* planned cardiac surgery,
* high risk of short-term non-cardiac death,
* planned management within rehabilitation center/HF clinic at discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with all cause death or unplanned hospitalization at 6 months | 6 months

SECONDARY OUTCOMES:
All cause mortality at 12 months | one year
Unplanned HF-related hospitalization at 6 and 12 months | 6 and 12 months
Number of alive and hospitalization-free days at 6 and 12 months | 6 and 12 months
Mean and distribution modified Goldman classe at 6 months | 6 months
Natriuretic peptides blood levels at 6 months. | 6 months.
Global cost of patient management | from day0 to 12 months
HF-treatment at 6 months | 6 months
Mean and distribution NYHA classe at 6 months | 6 months
Analysis of subgroups (LVEF altered or not, first HF episode or not, age> or ≤ 75, Changes in levels of BNP or NT-proBNP between day0 and the second consultation in the active group: ≥ 30% decrease, ≥ 30% increase, Intermediate variation). | 6 months
Biomarkers measured in plasma collected at day0: predictive value of the risk of death and hospitalization during the period of 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: LOGEART Damien, MD, PhD, Principal Investigator — Lariboisiere Hospital, APHP
Locations (1):
- Service de Cardiologie - Hopital Lariboisière, Paris, France